CLINICAL TRIAL: NCT05578664
Title: Efficacy of PErioperative PEmbrolizumab Treatment in Patients With Resectable Metastases From Kidney Cancer. (The PE-PE Study).
Brief Title: Efficacy of PErioperative PEmbrolizumab Treatment in Patients With Resectable Metastases From Kidney Cancer
Acronym: PE-PE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorzio Oncotech (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PE-PE
Record Dates: First submitted 2022-10-07; First posted 2022-10-13 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Oligometastatic Renal Cell Carcinoma
MeSH Terms: interventions — pembrolizumab; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups (ARM A vs ARM B) in parallel for the duration of the study.
  Eligible patients will be randomized 2:1 to receive:
  * ARM A: pembrolizumab at flat dose of 400 mg every six weeks for a total of 9 cycles (one year of therapy) and metastasis directed treatment (surgery or RT) from day 21 of cycle 1 to day 42 of cycle 1; OR
  * ARM B: local therapy alone within 42 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A (Experimental): Pembrolizumab will be administered at flat dose of 400 mg IV every six weeks for a total of 9 cycles (one year of therapy) and metastasis directed treatment (surgery or RadioTherapy, RT) from day 21 of cycle 1 to day 42 of cycle 1.
  Interventions: Drug: Pembrolizumab injection plus metastasis directed treatment (surgery or RT); Other: Tumor resection or RT
- ARM B (Active Comparator): Local therapy alone (tumor resection or definitive RadioTherapy, RT) within 42 days from randomization.
  Interventions: Other: Tumor resection or RT

INTERVENTIONS:
Drug: Pembrolizumab injection plus metastasis directed treatment (surgery or RT) — Pembrolizumab 400 mg will be administered as a 30 minute IV infusion every 6 weeks for a total of 9 cycles (one year of therapy) and metastasis directed treatment (surgery or RT) from day 21 of cycle 1 to day 42 of cycle 1
  Arms: ARM A
Other: Tumor resection or RT — Tumor resection or RT will be applied within 42 days from randomization.

SUMMARY:
This is a phase II trial aiming at assessing the efficacy of pembrolizumab to delay tumor progression in patients with oligometastatic clear cell metastatic Renal Cell Carcinoma (mRCC).

Eligible patients for this trial should have received previous surgery for primary tumor and have maximum of three metastases considered eligible for radical therapy (surgery or metastases directed radiotherapy).

Eligible patients will be randomized 2:1 to receive:

* ARM A: pembrolizumab at flat dose of 400 mg every six weeks for a total of 9 cycles (one year of therapy) and metastasis directed treatment (surgery or RT) from day 21 of cycle 1 to day 42 of cycle 1; or
* ARM B: local therapy alone within 42 days.

DETAILED DESCRIPTION:
In this study, approximately 81 participants with ccRCC will be enrolled. The RESORT and E2810 clinical trials reported a rate of patients free of relapse of about 50% at 24 months. This study aims to improve this rate from 50% to 70% corresponding to an Hard Ratio of 0.51. Therefore, the sample size required for demonstrating this relapse-free survival (RFS) advantage includes a total of 74 patients that will be randomized 2:1 in the arm A or B respectively. The study will detect a treatment difference with the 80% probability at a one-sided p and 10.0% significance level, if the true hazard ratio is 0.51. This is based on the assumption that the accrual period will be 30 months, the follow up period will be 24 months, and the median RFS is 24 months.

Because 10% of dropout has been estimated, the final number of patients is 81.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of clear cell renal cell carcinoma will be enrolled in this study.
2. Have undergone a partial nephrectomy or radical complete nephrectomy with negative surgical margins.
3. Evidence of oligo-metastatic disease eligible for local treatment with radiotherapy or surgery, defined as:

   1. Appearance of new metastases within 5 years from previous eradication of primary tumors or previous metastasectomy.
   2. Presence of maximum 3 metastases in the same site or in different sites with the exception of bone metastases that cannot exceed the number of 2 if they are the sole disease site or one in case of multiple sites.
   3. Each metastasis should be less than 3 cm in the maximum diameter and less than 5 cm in the sum of the longest tumor diameters (this evaluation should apply also for lymph nodes).
4. Has received no prior systemic therapy for Renal Cell Carcinoma (RCC).
5. Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 7 days of before the start of study intervention.
6. The participant (or legally acceptable representative) has provided documented informed consent/assent for the study.
7. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a primary tumor or tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slide. Newly obtained biopsies are preferred to archived tissue.

   Female participants:
8. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 of the Study protocol OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days (corresponding to time needed to eliminate any study treatment(s)) plus 30 days (a menstruation cycle) for study treatments with risk of genotoxicity after the last dose of study treatment.
9. Adequate organ function defined as:

System - Laboratory Value

Hematological

* Absolute neutrophil count (ANC): ≥ 1500/μl
* Platelets: ≥ 100 000/μl
* Hemoglobin: ≥ 9.0 g/dL or ≥ 5.6 mmol/L

Renal

* Creatinine: ≤1.5 x Upper Limit of Normal (ULN) OR
* Measured or calculated creatinine clearance: ≥ 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN (GFR can also be used in place of creatinine or CrCl)

Hepatic

* Total bilirubin: ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 x ULN
* Aspartate transaminase (AST or SGOT) and alanine transaminase (ALT or SGPT): ≤ 2.5 x ULN (≤ 5 ULN for participants with liver metastases)

Coagulation

* International normalized ratio (INR) OR prothrombin time (PT)
* Activated partial thromboplastin time (aPTT): ≤ 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

1. Has had major surgery, other than nephrectomy, within 4 weeks prior to randomization.

   Note: If participants received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
2. Has residual thrombus post nephrectomy in the vena renalis or vena cava.
3. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
4. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to randomization.

   Note: Participants must have recovered from all Adverse Events (AEs) due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible. Participants with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible
5. Has clinically significant cardiovascular disease within 12 months from first dose of study intervention, including NYHA Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, undergone CABG or PTCA, or cardiac arrhythmia.

   Note: Medically controlled arrhythmia stable on medication is permitted.
6. Has moderate to severe hepatic impairment (Child-Pugh B or C).
7. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
8. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
9. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
10. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
11. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, non-muscle invasive bladder cancer, prostate cancer pT2 or less, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
12. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously surgically treated brain metastases may participate provided they are not radiological evidence of disease at the time of screening and without evidence of progression for at least 12 months by repeat imaging (note that the repeat imaging should be performed during study screening).
13. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
14. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
15. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
16. Has an active infection requiring systemic therapy.
17. Has a known history of Human Immunodeficiency Virus (HIV) infection.
18. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (HCV, defined as HCV RNA is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
19. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
20. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
21. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
22. Has had an allogenic tissue/solid organ transplant.
23. A WOCBP who has a positive urine pregnancy test within 72 hours prior to randomization. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Relapsed Free Survival (RFS) | 24 months
  The length of time from the randomization and the appearance of radiological progression of kidney cancer in patients who received pembrolizumab compared to those who did not

SECONDARY OUTCOMES:
Distant Relapsed Free Survival (Distant RFS) | 24 months
  The length of time from the randomization to the appearance of distant metastases outside those treated with surgery or radiotherapy.
Overall Survival (OS) | 24 months
  The time from the randomization to the patient's death or last contact in patients who received pembrolizumab compared to those who did not.
Safety Endpoint | 24 months
  The overall incidence of adverse events in patients who received pembrolizumab compared to those who did not.
Local Progression Disease (Local PD) | 24 months
  The overall incidence local progression in patients who received pembrolizumab plus RT compared to those who received RT alone

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Iacovelli, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario "A. Gemelli" IRCCS - UOC Oncologia Medica, Rome
Locations (1):
- Fondazione Policlinico Universitario "A. Gemelli" IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No